CLINICAL TRIAL: NCT03838562
Title: Non-inferiority of Virtual Reality Compared to Other Forms of Optokinetic Stimulation in the Rehabilitation of Vestibular Syndromes. Randomized Controlled Trial.
Brief Title: Virtual Reality Compared to Other Forms of Optokinetic Stimulation in the Rehabilitation of Vestibular Syndromes.
Acronym: EquiRV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL18_0243; 2018-A02247-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-01-28; First posted 2019-02-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-04

CONDITIONS: Vestibular Syndrome; Optokinetic Stimulation
Keywords: virtual reality; vestibular; balance; rehabilitation
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Arm (Experimental)
  Interventions: Other: Vestibular rehabilitation with virtual reality
- Control Arm (Active Comparator)
  Interventions: Other: Standard optokinetic stimulator or dynamic visual surround

INTERVENTIONS:
Other: Vestibular rehabilitation with virtual reality — Both group follow three or four weeks of vestibular rehabilitation program with 2 sessions of physical therapy per day and one collective session of balance exercices per day, five day per week. More orthoptist care and muscle strengthening.
  The exercises performed include rotating exercises, static balance exercises with eyes open and closed, head fixed and with head oscillation. Exercises on unstable planes and on dynamic force platforms. Different walking and eye stabilization exercises.
  Only visual misinformation is distinct in both groups. Optokinetic application with three-dimensional head-mounted is used in the experimental group.
  Arms: Virtual Reality Arm
Other: Standard optokinetic stimulator or dynamic visual surround — Both group follow three or four weeks of vestibular rehabilitation program with 2 sessions of physical therapy per day and one collective session of balance exercices per day, five day per week. More orthoptist care and muscle strengthening.
  The exercises performed include rotating exercises, static balance exercises with eyes open and closed, head fixed and with head oscillation. Exercises on unstable planes and on dynamic force platforms. Different walking and eye stabilization exercises.
  Only visual misinformation is distinct in both groups. Standard optokinetic stimulator (stimulopt) or dynamic visual surround (smart equitest) are used in the control group.
  Arms: Control Arm

SUMMARY:
Context and justification: Vertigo leads to medical consultation, interruption of daily activities or work stoppage in 80% of cases. Optokinetic stimulation is used in awareness and adaptation exercises. The technology of three-dimensional head-mounted provides a strong immersion allowing optokinetic stimulation but studies interested in virtual reality in the context of balance rehabilitation have not been able to highlight the superiority of this therapy. The investigators therefore propose a non-inferiority trial because of the affordable price and small size of three-dimensional head-mounted.

Objectives : The objective of this study is to evaluate whether a rehabilitation program using virtual reality is as effective as a reference program using Smart Equitest and an optokinetic stimulator to improve the balance of patients with vestibular syndrome after 3 or 4 weeks of rehabilitation.

The investigators also assess the disability related to vertigo and balance disorders as well as the tolerance of virtual reality Methodology: Prospective, randomized controlled non-inferiority trial, monocentric, 2 parallel arm, with blind assessed after 3 or 4 weeks of follow-up.

The inclusion criteria are the pathologies eligible for a vestibular rehabilitation program and the possible standing position.

The criteria for non-inclusion are visually impaired or blind subjects, lack of relief vision, history of epilepsy, significant strabismus, permanent bilateral vestibular areflexes and Ménière's disease.

The main evaluation criterion is the balance score obtained with eyes closed on an unstable plane during a sensory organization test performed on a dynamic posturology platform, obtained during the final evaluation.

The secondary judgment criteria are:

* The balance scores obtained in the sensory organization test under other conditions.
* The Dizziness Handicap Inventory obtained during the final evaluation and three months after the end of the program.
* The tolerance of virtual reality will be measured weekly by the Simulator Sickness Questionnaire.

Statistics: The number of subjects to be included is 76, the analysis will first be performed per-protocol, the difference in scores between the two groups will be calculated, as well as its 95% confidence interval. If the lower bound of this interval is above the non-inferiority threshold, the same analysis will be performed on the population intending to treat (all randomized patients).

Process: Recruitment and rehabilitation take place at the CH Coste Floret. The duration of inclusions is 27 months, The duration of patient participation in the protocol is 4 months. Patients are cared for 21 or 28 days with two sessions of physiotherapy per day, five days a week, then resolved by telephone 3 months after the rehabilitation Feasibility: CH Coste Floret has the human and material resources necessary to carry out the protocol. The PMSI data show that the department receives about 40 patients per year who are likely to participate in the protocol.

Outcomes / perspectives: In the event of a result validating the non-inferiority of virtual reality, this study could provide further evidence of the value of this type of tool for the rehabilitation of subjects suffering from vestibular disorders. In addition, a medico-economic study would be possible in order to reinforce the advantages of virtual reality helmets.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatology related to a vestibular disorder, eligible for a rehabilitation program Possible standing position
* Informed subject and having signed the informed consent form
* Major subject
* Affiliation to a social security scheme

Exclusion Criteria:

* Badly sighted or blind subject (sharpness <1 / 10th)
* Absence of vision of the reliefs
* Strabismus important
* History of epilepsy
* General state strongly altered
* Pregnant subject
* Major protected by law
* Subject deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Balance score with eyes closed on an unstable plane during a sensory organization test | after 3 or 4 weeks of rehabilitation
  Realized with the Framiral® multitest equilibre. Framiral multitest equilibre is a posturography platform for performing vestibular assessments and targeted rehabilitation exercises

SECONDARY OUTCOMES:
Others score of the sensory organization test | 3 or 4 weeks
  Realized with the Framiral® multitest equilibre.Framiral multitest equilibre is a posturography platform for performing vestibular assessments and targeted rehabilitation exercises
The Dizziness Handicap Inventory | 3 or 4 weeks
The Dizziness Handicap Inventory | 4 month
The Simulator Sickness Questionnaire | weekly from week 1 to week 3 or 4
  This questionnaire includes the following questions: "Not at all", "A little", "Moderately" and "Severely", each answer is worth 0, 1, 2 or 3 points. The total score is equal to 48, the two scores are calculable "Nausea" on 27 and "Oculomotor" on 21. The higher the score, the more the side effects are important.l 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CH Paul Coste Floret/ Pavillon Jeanne d'Arc/ Leroy, Lamalou-les-Bains, France

REFERENCES:
- [Derived] Le Perf G, Thebault G, Duflos C, Herman F, Cauquil-Gleizes S, Laffont I. Can virtual reality replace conventional vestibular rehabilitation tools in multisensory balance exercises for vestibular disorders? A non-inferiority study. J Neuroeng Rehabil. 2025 Apr 19;22(1):86. doi: 10.1186/s12984-025-01623-x. PMID 40253374